CLINICAL TRIAL: NCT00544921
Title: Phase 1 Study of Anti-glycation Agent GLY-230
Brief Title: Phase 1 Study of Anti-glycation Agent GLY-230 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Glycadia (Industry)
Collaborators: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: GLY-001
Record Dates: First submitted 2007-10-15; First posted 2007-10-16 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — 2-(3-chlorophenylamino)phenylacetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- 50 mg (Experimental)
  Interventions: Drug: GLY-230
- 100 mg (Experimental)
  Interventions: Drug: GLY-230
- 250 mg (Experimental)
  Interventions: Drug: GLY-230
- 500 mg (Experimental)
  Interventions: Drug: GLY-230
- 750 mg (Experimental)
  Interventions: Drug: GLY-230
- 1000 mg (Experimental)
  Interventions: Drug: GLY-230
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GLY-230
  Arms: 100 mg; 1000 mg; 250 mg; 50 mg; 500 mg; 750 mg
Other: Placebo — No drug administered
  Arms: Placebo

SUMMARY:
To test the safety of GLY-230 and to evaluate how long drug stays in blood after taking it by mouth.

ELIGIBILITY:
Inclusion Criteria:

* Men age 18-55
* Negative drug screen
* Normal EKG, clinical chemistries, CBC, urinalysis, and
* Give written informed consent

Exclusion Criteria:

* Active concomitant serious medical or surgical disease,
* Hepatic or renal laboratory values above reference range, ise of other experimental drug within previous 30 days

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2005-10; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
A Dose-Ranging Study to Evaluate the Phamacokinetics and Safety of Six Single-Dose Levels of GLY-230 in Healthy Subjects | October, 2005 to October, 2006

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Kennedy, Principal Investigator — Univ. FLA Gainesville
Locations (1):
- Univ FL, Gainesville, Florida, United States